CLINICAL TRIAL: NCT00774956
Title: Shoulder Training: Muscle Recruitment Patterns and the Effect of an Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/432
Record Dates: First submitted 2008-09-25; First posted 2008-10-17 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subject with shoulder impingement
  Interventions: Procedure: Exercise training program
- 2 (Active Comparator): Healthy persons
  Interventions: Procedure: Exercise training program

INTERVENTIONS:
Procedure: Exercise training program — A 6 week shoulder exercise training program
  Arms: 1
Procedure: Exercise training program — A 6 week shoulder exercise training program
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the muscle recruitment pattern and the effect of a 6 week shoulder exercise training program in healthy persons and subjects with shoulder impingement

ELIGIBILITY:
Inclusion Criteria:

* current reported history of shoulder pain localised at the glenohumeral joint diagnosed as impingement
* two positive shoulder impingement tests
* pain reproduction during two of three additional categories of clinical tests
* the subject is able to perform pain-free arm elevations with a resistance of 0.5 kg

Exclusion Criteria:

* cervical and periscapular pain
* positive labral injury tests
* history of shoulder surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Muscle recruitment pattern | After 6 weeks of training

SECONDARY OUTCOMES:
Shoulder pain and functional ability in the patient group | After 6 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vanderstraeten, MD, PhD, Principal Investigator — University Ghent; Ann Cools, PhD, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium